CLINICAL TRIAL: NCT02429765
Title: Effect of Aclidinium Bromide/Formoterol on Nighttime Lung Function, Respiratory Mechanics and Early Morning Symptoms in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effect of Aclidinium/Formoterol on Nighttime Lung Function and Morning Symptoms in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMED-1744-14
Record Dates: First submitted 2014-11-07; First posted 2015-04-29 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACL/FOR (Active Comparator): The evening dose of twice-daily dual bronchodilator medication will consist of aclidinium/formoterol 400/12mcg . After 2-weeks of treatment with twice-daily aclidinium/formoterol 400/12mcg, subjects will be randomized to receive an evening dose consisting of active drug or placebo.
  Interventions: Drug: ACL/FOR
- Placebo (Placebo Comparator): The evening dose of twice-daily dual bronchodilator medication will consist of a placebo inhaler. After 2-weeks of treatment with twice-daily aclidinium/formoterol 400/12mcg, subjects will be randomized to receive an evening dose consisting of active drug or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACL/FOR
  Other Names: aclidinium/formoterol, Duaklir
  Arms: ACL/FOR
Drug: Placebo
  Arms: Placebo

SUMMARY:
A number of studies have documented poor sleep quality and troublesome symptoms (breathlessness, cough and sputum production) upon awakening in patients with COPD. However, the investigators know very little about measurements of respiratory mechanics (i.e., lung volumes, respiratory pressures, diaphragm function, etc) during sleep in these patients. The investigators also know little about how modern bronchodilator therapies, or the timing of when they are taken, affect respiratory mechanics during sleep or the severity of early morning respiratory symptoms. COPD is often treated with inhaled bronchodilator medications which are used to open up airways and make it easier for air to get in and out of the lungs. The investigators are studying the effects of a new inhaler that contains two different types of long-acting bronchodilator: formoterol [a long-acting beta2-agonist (LABA)] and aclidinium bromide [a long-acting muscarinic antagonist (LAMA) or anticholinergic]. Initial studies have shown that this combination therapy taken twice daily can improve some lung function measurements and respiratory symptoms in patients with moderate to severe COPD. There are also reports that evening administration of this medication may provide important advantages in patients with dominant nighttime and early morning symptoms. It is thought that sustained bronchodilation and lung deflation during the night may improve respiratory mechanics, diaphragmatic function, pulmonary gas exchange, sleep quality, and reduce severity of morning symptoms. This study will be the first to explore the effects of a nighttime dose of aclidinium/formoterol combination therapy on detailed measurements of respiratory mechanics and early morning symptoms in COPD. This study will also give us a better understanding of the mechanisms of early morning respiratory symptoms and their improvement with bronchodilators.

DETAILED DESCRIPTION:
STUDY DESIGN: This will be a randomized, placebo-controlled crossover study where patients will receive an evening dose of either aclidinium/formoterol (ACL/FOR) or placebo after steady-state conditions on twice-daily ACL/FOR have been established. Patients will continue to take the same dosage of inhaled corticosteroid (ICS) as they did prior to study entry. Subjects will complete 4 visits as part of the study, with a fifth follow-up visit if required to ensure return to pre-study health status. After an initial screening visit (Visit 1) to confirm eligibility and a 1-week run-in period on stable triple therapy [long-acting beta2-agonist/inhaled corticosteroid (LABA/ICS) + long-acting muscarinic antagonist (LAMA)], subjects will complete baseline testing (Visit 2) which includes: full pulmonary function tests, sleep/symptom questionnaires, and polysomnography which will include periodic measurements of overnight spirometry (sitting and supine). Subjects will then receive 2-week treatment with twice-daily ACL/FOR and continue on the same ICS as during the baseline run-in. Once stability on treatment with ACL/FOR and ICS is established, there will be two overnight treatment visits (Visits 3 and 4), conducted 3-7 days apart to allow for return to normal sleep status between. For these visits, the evening dose of ACL/FOR versus placebo will be randomized to treatment order. Treatment visits will be similar to visit 2 but will include overnight measurements of respiratory mechanics (diaphragm electromyography and respiratory pressures). Short-acting bronchodilators will be withheld for at least 8 hours prior to visits.

SAMPLE SIZE: This is an exploratory physiological study with the primary outcome being an improvement in morning pre-dose trough inspiratory capacity (IC) by 200 ml. A sample size of 20 will provide at least 80% to detect this treatment difference based on a standard deviation (SD) of approximately 0.2 L for a response difference in trough IC (vanNoord, 2006), a two-tailed test and a p<0.05. The investigators anticipate that all patients will not consent to instrumentation; however, the investigators are hoping for n=12 with respiratory mechanical measurements. Due to the complexity of the study and its measurements, an interim analysis will be conducted after 10 subjects have been completed.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe COPD (post-bronchodilator forced expiratory volume in 1 s (FEV1) 30-79%predicted);
* Resting functional residual capacity (FRC) >120% predicted;
* Clinically stable and on stable triple therapy with an ICS/LABA and tiotropium;
* Symptomatic: Baseline Dyspnea Index ≤8 and answer "in the morning" when asked about what time of day their COPD symptoms are worst.

Exclusion Criteria:

* A diagnosis of sleep disordered breathing;
* Nocturnal oxygen therapy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Morning trough inspiratory capacity (IC) as measured by a spirometer | 10 hours after the evening dose of randomized study drug
  Early morning IC (~6:00am) will be measured to assess improvements in lung hyperinflation in response to the evening dose (~8:00pm) of a twice-daily bronchodilator vs. placebo.

SECONDARY OUTCOMES:
Early Morning Symptoms of COPD Instrument (EMSCI) | Upon awakening in the morning: 10 hours after the evening dose of randomized study drug
Distribution of sleep stages obtained during polysomnography | Participants will be followed for the duration of the night after the evening dose of randomized study medication: between bedtime at 10pm and upon waking or 5:45am, whichever is sooner
Changes in the forced expired volume in 1 second (FEV1) as measured by a spirometer | Measurements will be collected at 2-hr intervals after the evening dose of randomized study medication (i.e., 2, 4, 6, 8 and 10 hrs post-dose)
Changes in IC as measured by a spirometer | Measurements will be collected at 2-hr intervals after the evening dose of randomized study medication (i.e., 2, 4, 6, 8 and 10 hrs post-dose)
Morning trough functional residual capacity (FRC) as measured by body plethysmography | 10 hours after the evening dose of randomized study drug
  For assessment of lung hyperinflation
Diaphragm electromyography (EMGdi) | Measurements will be collected at 2-hr intervals after the evening dose of randomized study medication (i.e., 2, 4, 6, 8 and 10 hrs post-dose)
  A combined electrode-balloon esophageal/gastric catheter will be inserted nasally to measure EMGdi and respiratory pressures (esophageal and gastric pressures)
Transdiaphragmatic pressure (Pdi) | Measurements will be collected at 2-hr intervals after the evening dose of randomized study medication (i.e., 2, 4, 6, 8 and 10 hrs post-dose)
  A combined electrode-balloon esophageal/gastric catheter will be inserted nasally to measure EMGdi and respiratory pressures (esophageal and gastric pressures). Transdiaphragmatic pressure is calculated as the difference between esophageal pressure and gastric pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University & Kingston General Hospital
Locations (1):
- Respiratory Investigation Unit, Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Domnik NJ, Phillips DB, James MD, Ayoo GA, Taylor SM, Scheeren RE, Di Luch AT, Milne KM, Vincent SG, Elbehairy AF, Crinion SJ, Driver HS, Neder JA, O'Donnell DE. Compensatory responses to increased mechanical abnormalities in COPD during sleep. Eur J Appl Physiol. 2022 Mar;122(3):663-676. doi: 10.1007/s00421-021-04869-0. Epub 2022 Jan 16. PMID 35034195
- [Derived] Domnik NJ, James MD, Scheeren RE, Ayoo GA, Taylor SM, Di Luch AT, Milne KM, Vincent SG, Phillips DB, Elbehairy AF, Crinion SJ, Driver HS, Neder JA, O'Donnell DE. Deterioration of Nighttime Respiratory Mechanics in COPD: Impact of Bronchodilator Therapy. Chest. 2021 Jan;159(1):116-127. doi: 10.1016/j.chest.2020.06.033. Epub 2020 Jun 27. PMID 32603714